CLINICAL TRIAL: NCT06227676
Title: Formative Assessment of the Effect of 'Cramp Bites' Intake on Primary Dysmenorrhea in Women Aged 18-25: A Placebo-Controlled Trial
Brief Title: Effect of 'Cramp Bites' on Period Cramps in Women Aged 18-25
Acronym: NUTRITION; GYN
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cornell University (Other)
Collaborators: Laidlaw Foundation (Unknown); Epperson Fund (Unknown); Beck Fellowship (Unknown); Dan Cane Fund (Unknown)
Responsible Party: Principal Investigator, Armita Jamshidi, Women's Health Student, Cornell University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB0145243
Record Dates: First submitted 2024-01-17; First posted 2024-01-29 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Dysmenorrhea Primary; Dysmenorrhea; Menstrual Discomfort; Menstrual Problem; Menstrual Cycle Abnormal; Menstrual Pain; Period Pain; Period Problem; PMS; Premenstrual Syndrome; PCOS; PCOS (Polycystic Ovary Syndrome) of Bilateral Ovaries; PCOS (Polycystic Ovary Syndrome) of Left Ovary; PCOS (Polycystic Ovary Syndrome) of Right Ovary; Polycystic Ovary Syndrome; Premenstrual Dysphoric Disorder; Cramps; Ovarian Cysts
Keywords: Dysmenorrhea; Primary Dysmenorrhea; Menstrual Discomfort; Menstrual Pain; Menstrual Problem; Menstrual Cycle Abnormal; Period Pain; Period Problem; PMS; Premenstrual Syndrome; PCOS; PCOS (Polycystic Ovary Syndrome) of Bilateral Ovaries; PCOS (Polycystic Ovary Syndrome) of Left Ovary; PCOS (Polycystic Ovary Syndrome) of Right Ovary; Polycystic Ovary Syndrome; Premenstrual Dysphoric Disorder; Cramps; Ovarian Cysts
MeSH Terms: conditions — Dysmenorrhea; Menstruation Disturbances; Premenstrual Syndrome; Polycystic Ovary Syndrome; Premenstrual Dysphoric Disorder; Muscle Cramp; Ovarian Cysts

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned either 'Cramp Bites' or our Placebo Snack over the duration of one menstrual cycle.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Granola Bites (Placebo Comparator): This snack contains no known spices or nutrients that have been shown to help with spasmodic or congestive dysmenorrhea. It is the same shape and size as the active comparator.
  Interventions: Dietary Supplement: Cramp Bites by Aunt Flo's Kitchen
- Cramp Bites (Active Comparator): This snack contains spices and ingredients that have been shown to help with both spasmodic and congestive dysmenorrhea. It is the same shape and size as the placebo comparator.
  Interventions: Dietary Supplement: Cramp Bites by Aunt Flo's Kitchen

INTERVENTIONS:
Dietary Supplement: Cramp Bites by Aunt Flo's Kitchen — Participants who are randomly assigned this snack are instructed to eat one serving each day, starting 2 days before their next onset of menstruation, and extending 3 days into their menstrual cycle. They are instructed to eat their assigned snack each time they experience menstrual cramps, whether spasmodic or congestive.
  Other Names: Aunt Flo's Kitchen; SheBalls LLC; Period Snack; Natural Period Snack; Armita Jamshidi; Period Cramp Food; Menstrual Cramp Food; Menstrual Cramp Alleviant; Period Pain Food; Menstrual Pain Food; Natural Period Cramp; Natural Menstrual Cramp

SUMMARY:
85 percent of women of reproductive age experience consistent period cramps/menstrual pain, and 60% indicate that they do not use painkillers to relieve menstrual symptoms; there is a need for natural and non-medicative supplements to dysmenorrhea. The purpose of this clinical trial is to examine the effect of 'Cramp Bites'--classified by a mixture of natural ingredients researched to help with period pain--on women suffering from primary dysmenorrhea: this will be done through providing participants with the snack and surveying them on how it changes their period symptoms.

DETAILED DESCRIPTION:
Participants will be asked the following information at the interview: name, month and year of birth, ethnicity, email, and phone number. As well, they will be prompted for their lifestyle habits, allergies, prior pregnancies and deliveries, presence of pathological disorders, medication (specifically asking about oral contraception), use of over-the-counter painkillers for period cramps/menstrual pain, expected date of next period, and menstrual cycle history. They will also be asked to complete the Menstrual Symptom Questionnaire.

The baseline questionnaire will ask the participant about their prior experience with primary dysmenorrhea symptoms and with period cramps/menstrual pain on a sliding scale.

The daily questionnaire will ask the participant to rate the extent of their period cramps/menstrual pain, to describe their pain, and whether they have taken any drugs for their period pain on that day. This questionnaire will be completed by all participants starting 2 days before their next onset of menstruation. Participants were randomly assigned Cramp Bites or the Placebo Snack: all other protocols remain the same.

After their next menstrual cycle ends, participants will be asked to fill out a final questionnaire: this questionnaire will ask the participant if they have noticed any changes in their period pain, the efficacy of the snack, and if they have suggestions/comments about the snack. This study is divided into 4 parts. Some parts will take place at Cornell University, and other parts can be completed online.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18 and 25 who experience primary dysmenorrhea and have no pathological disorders.

Exclusion Criteria:

* Pregnancy or breast feeding within 6 months
* Primary or secondary amenorrhea
* Body mass index less than the 1st percentile or body weight above 300 lbs
* Undergoing menstrual suppression by medicative means
* Unwilling to avoid painkillers (ibuprofen or naproxen) for the duration of the study unless absolutely necessary
* Has allergies or aversions to ingredients used in either Cramp Bites or the Placebo Snack
* Not fluent in English

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants must be assigned female at birth to be eligible for the study.
Enrollment: 12 (Actual)
Dates: Start 2022-07-21 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale for Spasmodic Cramps | Participants complete this survey when they experience cramps: once before they consume their snack, and once after. Completion time for each survey is 7 minutes.
  Participants rate their spasmodic cramp severity before and after eating either Cramp Bites or the Placebo Snack using the Visual Analogue Scale. This is on a scale from 0 to 10, where 0 represents no cramps and 10 indicates extreme abdominal cramping.
Visual Analogue Scale for Congestive Cramps | Participants complete this survey when they experience cramps: once before they consume their snack, and once after. Completion time for each survey is 7 minutes.
  Participants rate their congestive cramp severity before and after eating either Cramp Bites or the Placebo Snack using the Visual Analogue Scale. This is on a scale from 0 to 10, where 0 represents no cramps and 10 indicates extreme abdominal cramping.

SECONDARY OUTCOMES:
Menstrual Symptom Questionnaire (MSQ) | Participants complete this questionnaire with a researcher before the study. Time to complete this questionnaire is 15 minutes.
  Filled out during intake exam. MSQ indicates to what extent the participant suffers from spasmodic cramps, congestive cramps, or a mixture of the two.

OTHER OUTCOMES:
Product Feedback Form | Participants were asked to fill out this survey at the end of the study. Completion time was 5 minutes.
  Participants are asked to fill out a feedback form indicating how confident they were about their assigned snack's efficacy and the taste of the snack.

CONTACTS AND LOCATIONS:
Locations (1):
- Cornell University, Ithaca, New York, United States

IPD SHARING:
Plan to Share IPD: No
Due to the privacy protection of participants, individual participant data will not be disclosed.

REFERENCES:
- [Background] Iacovides S, Avidon I, Baker FC. What we know about primary dysmenorrhea today: a critical review. Hum Reprod Update. 2015 Nov-Dec;21(6):762-78. doi: 10.1093/humupd/dmv039. Epub 2015 Sep 7. PMID 26346058
- [Background] Ferries-Rowe E, Corey E, Archer JS. Primary Dysmenorrhea: Diagnosis and Therapy. Obstet Gynecol. 2020 Nov;136(5):1047-1058. doi: 10.1097/AOG.0000000000004096. PMID 33030880
- [Background] Itani R, Soubra L, Karout S, Rahme D, Karout L, Khojah HMJ. Primary Dysmenorrhea: Pathophysiology, Diagnosis, and Treatment Updates. Korean J Fam Med. 2022 Mar;43(2):101-108. doi: 10.4082/kjfm.21.0103. Epub 2022 Mar 17. PMID 35320895
- [Background] Chen CX, Kwekkeboom KL, Ward SE. Self-report pain and symptom measures for primary dysmenorrhoea: a critical review. Eur J Pain. 2015 Mar;19(3):377-91. doi: 10.1002/ejp.556. PMID 25059384
- [Background] Chesney MA, Tasto DL. The development of the menstrual symptom questionnaire. Behav Res Ther. 1975 Oct;13(4):237-44. doi: 10.1016/0005-7967(75)90028-5. No abstract available. PMID 1238078
- [Background] Guimaraes I, Povoa AM. Primary Dysmenorrhea: Assessment and Treatment. Rev Bras Ginecol Obstet. 2020 Aug;42(8):501-507. doi: 10.1055/s-0040-1712131. Epub 2020 Jun 19. PMID 32559803
- [Background] Direkvand-Moghadam A, Khosravi A. The impact of a novel herbal Shirazi Thymus Vulgaris on primary dysmenorrhea in comparison to the classical chemical Ibuprofen. J Res Med Sci. 2012 Jul;17(7):668-70. PMID 23798928
- [Background] Mates L, Popa DS, Rusu ME, Fizesan I, Leucuta D. Walnut Intake Interventions Targeting Biomarkers of Metabolic Syndrome and Inflammation in Middle-Aged and Older Adults: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Antioxidants (Basel). 2022 Jul 21;11(7):1412. doi: 10.3390/antiox11071412. PMID 35883903
- [Background] Gutman G, Nunez AT, Fisher M. Dysmenorrhea in adolescents. Curr Probl Pediatr Adolesc Health Care. 2022 May;52(5):101186. doi: 10.1016/j.cppeds.2022.101186. Epub 2022 May 4. PMID 35523674
- [Background] Negriff S, Dorn LD, Hillman JB, Huang B. The measurement of menstrual symptoms: factor structure of the menstrual symptom questionnaire in adolescent girls. J Health Psychol. 2009 Oct;14(7):899-908. doi: 10.1177/1359105309340995. PMID 19786516